CLINICAL TRIAL: NCT01067560
Title: Measurement of CSF Glucose Levels Using Three Different Glucose Meters in Parturients Undergoing Spinal Anesthesia for Elective Cesarean Section
Brief Title: Measuring Cerebrospinal Fluid (CSF) Glucose Levels in Patients Under Going an Elective Cesarean Section With Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Giselle Villar, University of British Columbia
Other Study IDs: H09-02574
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Anesthesia
Keywords: Glucose; CSF; Cesarean section, spinal anesthesia; Nova Stat Strip; Abbott Precision Xtra; Roche Accucheck Inform 2

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, CSF
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will determine the level of glucose (sugar) in the CSF (fluid that surrounds the spinal cord) in 30 subjects having spinal anesthesia for cesarean section using a bedside glucose meter. Spinal anesthesia is done by injecting drugs through a needle into the CSF. Subjects will have 1/10 tsp of CSF removed at the time of spinal anesthesia to measure the level of glucose. Glucose meters measure glucose, usually in the blood, and they can be used in the operating room. This study will see whether a glucose meter will easily measure the level of glucose in CSF.

DETAILED DESCRIPTION:
Detailed Description Spinal anesthesia consists of putting drugs into the cerebrospinal fluid (CSF), the fluid that surrounds the spinal cord. This allows the subject to be awake but "numb" from the chest down during your operation. Spinal anesthesia is done by inserting a small needle (spinal needle) in the subject's back into the space (subarachnoid space) containing the CSF. Once the spinal needle is in the subarachnoid space a small amount of fluid (CSF) is seen coming out of the spinal needle, confirming that the needle is in the right space. The anesthesiologist then injects local anesthetic into the CSF to freeze or numb the area for your surgery and some pain medication, such as morphine, to relieve pain after the operation.

CSF contains glucose (sugar) and the presence of glucose in the fluid that comes out of a spinal needle will confirm that the fluid is CSF. If spinal anesthesia is used for cesarean section following failed epidural anesthesia (may happen in women who had an epidural for labor pain relief who then need a cesarean section) it may be difficult to tell whether the fluid that comes out of the spinal needle is CSF or local anesthetic used for the epidural. In other words, the needle may be in the epidural space instead of the subarachnoid space and so the spinal anesthetic would not work. A simple bedside test to confirm that the fluid is CSF could potentially prevent this situation. Local anesthetic does not contain glucose so testing the fluid for glucose could help determine if the needle is in the proper space for spinal anesthesia.

The study will determine the normal levels of CSF glucose using three different glucose meters (Nova Stat Strip, Abbott Precision Xtra and Roche Accucheck Inform 2 which are bedside devices that measure glucose). A glucose meter is used by people with diabetes to check their blood sugar levels using a drop of their blood. The results of this study will hopefully provide the basis for a further study that would look at whether it is possible to distinguish CSF from epidural fluid when spinal anesthesia is done following a failed epidural anesthetic. This could help prevent failures of spinal anesthesia in that situation.

This is a prospective, observational study.

The Cesarean Section and spinal anesthesia will continue as per usual practice at BCWH. Consenting subjects will receive the same drugs and all aspects of the anesthetic care will be the same except for two differences. The first, is that the anesthesiologist will collect a very small amount of CSF (0.5 mL which is 1/10 of a teaspoon) to measure the amount of glucose. This testing will be done in the operating room with the three glucose meters (Nova Stat Strip, Abbott Precision Xtra and Roche Accucheck Inform 2) and in the laboratory (using one of the two machines: 1)Vitros 9 or 2)Vitros 5,1 FS). Secondly, blood sugar level will be tested by taking up to three drops of blood from a pinprick in the subject's toe to compare with the CSF glucose level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (American Society of Anesthesiologists (ASA) 1 or 2 classification) with a singleton pregnancy who are undergoing Cesarean section under spinal anesthesia.
* Age 19 years or older
* Understand written and oral English

Exclusion Criteria:

* Women who are having an emergency Cesarean section
* Women who are having epidural, combined spinal epidural or general anesthesia
* Women who have a contraindication to spinal anesthesia
* Women who are less than 19 years of age
* Women with an abnormality of glucose metabolism such as diabetes mellitus, gestational diabetes
* Women receiving dextrose intravenously prior to their surgery
* Women in whom technical problems are anticipated during insertion of the spinal (such as scoliosis) ot who may have a hematological abnormality o If there is technical difficulty during insertion of the spinal there is an increased chance of trauma, resulting in blood entering the CSF (bloody tap). This could potentially be a source of glucose. Women with a hematological abnormality are at increased of bleeding which may increase the chance of blood in the CSF.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients undergoing Cesarean delivery under spinal anesthesia at BC Women's Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcome is to establish reference ranges for glucose in CSF in parturients undergoing Cesarean delivery under spinal anesthesia using glucose meters currently undergoing testing at BC Women's Hospital | 1 day

SECONDARY OUTCOMES:
Our secondary objective is to compare the performance of glucose meters (bed side testing devices for glucose) to measure CSF glucose via three glucose meters (Nova Stat Strip, Abbott Precision Xtra and Roche Accucheck Inform 2). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Villar, MD, Principal Investigator — University of British Columbia; Anne Catherine Halstead, MD, FRCPC, Study Director — University of British Columbia; Simrat Saran, MD, BSc, Study Director — University of British Columbia; Steve Thomas, MBChB, FRCA, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital, Department of Anesthesia, Vancouver, British Columbia, Canada